CLINICAL TRIAL: NCT06965153
Title: Peer Recovery Coaching for Promoting Tobacco Abstinence in People With Opioid Use Disorder
Brief Title: Peer Recovery Coaching for Tobacco Abstinence in People With Opioid Use Disorder
Acronym: PeerTTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joanna M. Streck, Ph.D., Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025P001024
Record Dates: First submitted 2025-05-01; First posted 2025-05-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Peer Recovery Coaching for TUD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PeerTTS (Experimental): Peer recovery coach-delivered tobacco cessation coaching plus dual NRT
  Interventions: Drug: Dual NRT; Behavioral: PeerTTS
- SOC (Active Comparator): Non-peer delivered tobacco cessation coaching plus dual NRT
  Interventions: Drug: Dual NRT

INTERVENTIONS:
Drug: Dual NRT — Dual nicotine replacement therapy
Behavioral: PeerTTS — Peer recovery coach delivered tobacco cessation coaching
  Arms: PeerTTS

SUMMARY:
Tobacco use is a leading cause of premature death among individuals with opioid use disorder (OUD). Nearly 75% of individuals receiving medication treatment for OUD report concurrent tobacco use disorder (MOUD-TUD), yet evidence-based TUD treatment (i.e., Food and Drug Administration-approved medications and counseling) is less effective in those with MOUD-TUD compared to the general smoking population. Innovative interventions for promoting TUD cessation in individuals with MOUD-TUD are urgently needed. Major factors maintaining TUD in those with OUD that have not been addressed in existing treatment interventions in this population are the small social networks comprised of other smokers, pro-smoking social norms in social networks, and limited social support for quitting smoking. Peer recovery coaches (PRCs) are people with lived OUD experience who provide peer coaching to individuals with OUD and have been shown to promote increased OUD treatment retention and illicit opioid abstinence. PRCs who are in OUD-TUD recovery and trained in TUD treatment, are well positioned to provide a social model for nonsmoking and to alter the pro-smoking social norms that maintain TUD in those receiving MOUD; but this has never been tested. The investigators hypothesize that a tobacco cessation intervention, delivered by PRCs in OUD and TUD recovery with TUD training, combined with a safe and effective FDA-approved cessation medication (dual nicotine replacement therapy [NRT]), will be feasible, acceptable and have a greater effect on tobacco abstinence rates than current standard care TUD treatment (non-peer delivered TUD coaching plus dual NRT). To test this hypothesis, in this 3-year pilot R34, the investigators propose to adapt a behavioral TUD intervention, PeerTTS, to people with OUD and TUD and to train PRCs in OUD and TUD recovery to deliver the intervention. The investigative team will then conduct a pilot randomized controlled trial (RCT) in 60 participants with MOUD-TUD interested in reducing or quitting tobacco at MGH. Participants will be randomized to receive 12 weeks of 1) PeerTTS, defined as PRC-delivered tobacco cessation coaching plus dual NRT or 2) standard care (SOC), defined as non-peer delivered TUD coaching plus dual NRT. The proposed work will adapt and test whether a peer recovery coach-delivered tobacco cessation intervention is feasible, acceptable, and potentially more effective than standard care, when combined with first line pharmacotherapy in those with MOUD-TUD. The pilot RCT will provide quantitative and qualitative data to inform a fully powered R01 or equivalent testing a refined version of the PeerTTS intervention for individuals with MOUD-TUD who face a disproportionate burden of tobacco use and related mortality. This proposal aligns with NIDA's high priority research areas to test novel treatments that sustain recovery in individuals with poly-substance use (OUD and TUD) and to advance the science of peer recovery support. It also aligns with calls to enhance PRC training to include additional evidence-based competencies that improve health.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years of age)
* reporting current daily cigarette smoking (≥ 5 cigarettes per day in past 7 days),
* who are interested in quitting or cutting down on smoking in the next 3 months (yes/no),
* stable on their medication treatment for OUD (MOUD) at MGH (confirmed with patient's buprenorphine prescriber).

Exclusion Criteria:

* life expectancies < 1 year (per chart review by physician Co-I) or with any serious psychiatric or cognitive problem that would preclude ability to provide informed consent (i.e., unstable or untreated bipolar disorder, schizophrenia spectrum disorder, psychotic disorder, or actively suicidal)
* participants who have recent unstable cardiovascular or cerebrovascular disease (e.g., recovery phase of acute myocardial infarction, severe cardiac arrhythmias, and cerebrovascular accident; See Human Subjects) per discussion with their MOUD prescriber.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility-PeerTTS session attendance | Baseline through 3 months
  PeerTTS coaching session attendance

SECONDARY OUTCOMES:
Biochemically confirmed past 7-day tobacco abstinence | 3 months
  CO-confirmed abstinence
Acceptability | 3 months
  Client Satisfaction Questionnaire (CSQ-8)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna M Streck, PhD, Principal Investigator — Massachusetts General Hospital